CLINICAL TRIAL: NCT00235261
Title: Effect of Paracetamol Versus Paracetamol Combined With Pregabalin Versus Paracetamol Combined With Pregabalin and Dexamethasone on Pain and Opioid Requirements in Patients Scheduled for a Primary Total Hip Replacement
Brief Title: Effect of Paracetamol, Pregabalin and Dexamethasone on Pain and Opioid Requirements in Patients After Hip Operations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SM3-05
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2007-08-17 (Estimated); Status verified 2007-08

CONDITIONS: Pain; Postoperative
Keywords: Total hip replacement; Pregablin; Dexamethasone; Multimodal postoperative analgesia.
MeSH Terms: conditions — Pain | interventions — Pregabalin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Pregabalin
Drug: Dexamethasone

SUMMARY:
Patients scheduled for primary total hip replacement needs postoperative pain treatment: i.e. morphine. Unfortunately morphine has side-effects: nausea, vomiting, sedation and dizziness, which is unpleasant for the patients and sometimes keeps them at bed longer time than needed. We investigate in new combinations of analgesics for postoperative pain, hoping to minimize the need for morphine and improve the patients pain score after operation.

DETAILED DESCRIPTION:
We investigate the effect of paracetamol versus paracetamol + pregabalin versus paracetamol + pregabalin + dexamethasone on pain and morphine usage in the first 24 hours postoperatively in patients getting a new hip alloplastic.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for primary total hip replacement in spinal anaesthesia
* between the age of 55 and 75,
* ASA 1-3, and with
* BMI between 18 and 35.

Exclusion Criteria:

* are unable to cooperate;
* does not speak Danish;
* has allergy for drugs used in the trial;
* has drug and/or medicine abuse;
* epilepsy;
* diabetes treated with medicine;
* treatment with systemic steroids within 4 weeks prior to the operation;
* daily use of antacids;
* daily use of analgesics except for NSAID, Cox2 inhibitors and Paracetamol;
* known kidney disease;
* use of antidepressants

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-10; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The total amount of morphine needed postoperatively from 0-4 h, and 0-24 h, administered by a patient controlled pain treatment. (PCA)

SECONDARY OUTCOMES:
Pain score (VAS) at rest and at mobilisation.
Postoperative nausea and vomiting.
Sedation.
Dizziness
All measurements are taken at 2,4 and 24 h postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Ole Mathiesen, MD, Study Chair — Department of Anaesthesiology, Copenhagen University Hospital in Glostrup, 2600 Glostrup, Denmark; Lars Steen Jacobsen, MD, Principal Investigator — Departmentof Anaesthesiology; Hørsholm Sygehus; Usserød Kongevej 102; 2970 Hørsholm; Denmark
Locations (1):
- Department of anaesthesiology; Hoersholm Sygehus, Hoersholm, Frederiksborg Amt, Denmark